CLINICAL TRIAL: NCT04622332
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study to Assess Safety and Efficacy of SIR1-365 in Patients With Severe COVID-19
Brief Title: A Pilot Study to Assess Safety and Efficacy of SIR1-365 in Patients With Severe COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sironax USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIR365-US-101
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SIR1-365 (Experimental): SIR1-365 dose 1 daily for 14 days
  Interventions: Drug: SIR1-365
- Matching placebo (Placebo Comparator): Matching placebo dose 1 daily for 14 days
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: SIR1-365 — Route of administration: oral
  Other Names: Pharmaceutical form: tablets
  Arms: SIR1-365
Drug: Matching Placebo — Route of administration: oral
  Other Names: Pharmaceutical form: tablets
  Arms: Matching placebo

SUMMARY:
Primary Objective:

• To evaluate overall safety and tolerability of SIR1-365 in patients with severe COVID-19

Secondary Objectives:

* To assess the clinical efficacy of SIR1-365 in patients with severe COVID-19
* To assess the effects of SIR1-365 on multiple inflammatory biomarker levels including C-reactive protein (CRP), ferritin, lymphocyte and neutrophil counts, cytokines, and chemokines
* To assess the effects of SIR1-365 on biomarkers indicative of target engagement in patients with severe COVID-19
* To assess the effects of SIR1-365 on biomarkers indicative of kidney injury in patients with severe COVID-19
* To assess the effects of SIR1-365 on biomarkers indicative of cardiovascular endothelial cell damage in patients with severe COVID-19
* To characterize plasma pharmacokinetics (PK) of SIR1-365 in patients with severe COVID-19

DETAILED DESCRIPTION:
Study duration per participant is approximately 28 days including a 14-day treatment period

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient with clinical diagnosis of SARS-CoV-2 virus infection per World Health Organization criteria including positive nucleic acid test of any specimen (e.g., respiratory, blood, or other bodily fluid) within 2 weeks prior to screening.
* Symptoms suggestive of severe systemic illness with COVID-19, which could include any of the following symptoms: fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, or shortness of breath at rest, or respiratory distress.
* Clinical signs indicative of severe systemic illness with COVID-19, which could include any of the following clinical signs: respiratory rate ≥ 30 per minutes, heart rate ≥ 125 per minute, SpO2 ≤ 93% on room air, or PaO2/FiO2 ratio < 300 mmHg.
* Men or women ≥18 but ≤80 years of age at the time of signing the informed consent.
* Patient is able to understand the purpose and risks of the study and provide signed and dated informed consent or have a legal representative provide consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

* Patient requires endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, extracorporeal membrane oxygenation (ECMO), or clinical diagnosis of respiratory failure.
* Patient with shock defined by systolic blood pressure < 90 mm Hg, or diastolic blood pressure < 60 mm Hg or requiring vasopressor.
* Patient with multi-organ dysfunction or failure defined by an increase in the Sequential Organ Failure Assessment score of 2 points or more.
* Patient is unlikely to survive beyond 2 days at the discretion of Investigator.
* Patient has used chronic systemic corticosteroids within 2 weeks prior to screening.
* Patient with positive results for human immunodeficiency virus (HIV) or hepatitis B or C test.
* Patient has known active tuberculosis (TB), history of uncontrolled TB, suspected or known systemic bacterial or fungal infections within 4 weeks prior to screening.
* Patient has any other condition, which makes the patient unsuitable for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Qu, Study Director — Sironax USA, Inc.
Locations (9):
- United States (3):
  - Triple O Research Institute, West Palm Beach, Florida
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Baptist Medical Center, Jackson, Mississippi
- Mexico (3):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Media Sur - Medica Sur Tlalpan, Tlalpan, Mexico City
  - Hospital Universitario "Dr. José Eleuterio González", Monterrey, Nuevo León
- Pakistan (3):
  - Dow University Hospital, Ojha Karachi, Karachi, Sindh
  - Sindh Infectious Disease Hospital, Karachi, Sindh
  - Aga Khan University Hospital, Karachi, Sindh

REFERENCES:
- [Derived] Chavez-Tapia N, Sayeed MA, Luxmi S, Kasper DJ, Xue F, Shen Y, Fan W, Yuan W, Du B. Safety and efficacy of selective RIPK1 inhibitor SIR1-365 in hospitalized patients with severe COVID-19: A multicenter, randomized, double-blind, phase 1b trial. J Intensive Med. 2024 Sep 12;5(1):70-78. doi: 10.1016/j.jointm.2024.07.003. eCollection 2025 Jan. PMID 39872839

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SIR1-365 | Matching placebo
Started | 24 | 21
Completed | 19 | 15
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Total: Total of all reporting groups
Arm/Group | SIR1-365 | Matching Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Categorical [Count of Participants; unit: Participants] — Population: Demographics is based on safety set
  Participants
    Age: <=18 years | 0 | 0 | 0
    Age: Between 18 and 65 years | 18 | 16 | 34
    Age: >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 11 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 6 | 14
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 3 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11
  Mexico | 10 | 11 | 21
  Pakistan | 6 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.75 (6.920) | 30.76 (6.786) | 30.20 (6.795)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Any TEAEs During the Treatment Period Baseline to Day 14
Description: Number of participants who experienced at least one treatment-emergent adverse event (TEAE), defined as any adverse event with an onset date on or after the first dose of study drug and up to and including Day 14 post-baseline, regardless of causality. TEAEs are reported per standard MedDRA terminology and severity grading. This is a safety endpoint assessed in the safety population.
Time Frame: Baseline to Day 14
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 5 | 10

2. Secondary Outcome: Secondary Safety Endpoint - 1 : Number of Patients With Any TEAEs During the Treatment Period Baseline to Day 28
Description: This secondary safety endpoint assesses the overall tolerability of the study intervention by counting the number of participants who experienced one or more treatment-emergent adverse events (TEAEs) during the specified treatment period
Time Frame: Baseline to Day 28
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 7 | 11

3. Secondary Outcome: Secondary Safety Endpoint -2 : Proportion of Patients With Any SAEs During the Study Baseline to Day 14
Description: This secondary safety endpoint evaluates the proportion of patients in the study population who experienced one or more serious adverse events (SAEs), as defined by regulatory standards (e.g., resulting in death, life-threatening events, hospitalization, persistent disability, or other medically significant conditions), occurring from baseline (Day 0) through Day 14 (inclusive)
Time Frame: Baseline to Day 14
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 1 | 5

4. Secondary Outcome: Secondary Safety Endpoint -3 : Number of Patients With Any SAEs During the Study Baseline to Day 28
Description: This secondary safety endpoint evaluates the proportion of patients in the study population who experienced one or more serious adverse events (SAEs), as defined by regulatory standards (e.g., resulting in death, life-threatening events, hospitalization, persistent disability, or other medically significant conditions), occurring from baseline (Day 0) through Day 28 (inclusive)
Time Frame: Baseline to Day 28
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 3 | 5

5. Secondary Outcome: Secondary Safety Endpoint -4 : Number of Patients With Any Drug-Related TEAE During the Study Baseline to Day 14
Description: This secondary safety endpoint assesses the incidence of any TEAE deemed related to the study drug (investigator-assessed causality) from baseline (Day 1, pre-dose) through Day 14 (inclusive). TEAEs are defined as adverse events (AEs) with an onset date on or after the first dose of study drug, regardless of severity or seriousness
Time Frame: Baseline to Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 2 | 1

6. Secondary Outcome: Secondary Safety Endpoint -5 : Number of Patients With Any Drug-Related TEAE During the Study Baseline to Day 28
Description: This secondary safety endpoint assesses the incidence of any TEAE deemed related to the study drug (investigator-assessed causality) from baseline (Day 1, pre-dose) through Day 28 (inclusive). TEAEs are defined as adverse events (AEs) with an onset date on or after the first dose of study drug, regardless of severity or seriousness
Time Frame: Baseline to Day 28
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Participants | 2 | 1

7. Secondary Outcome: Secondary Efficacy Endpoint -1 : Change in Derived PaO2/FiO2 Ratio From Baseline
Description: The PaO2/FiO2 ratio is a clinical measure of oxygenation efficiency, calculated as the arterial partial pressure of oxygen (PaO2, in mmHg) divided by the fraction of inspired oxygen (FiO2, expressed as a decimal between 0 and 1). The endpoint assesses the absolute change in this ratio from baseline (defined as the value at randomization or study entry, typically within 24 hours prior to intervention) to the specified post-baseline time point(s) (e.g., Day 7, End of Treatment, or as per protocol)
Time Frame: Baseline to EOT(Day 14)
Population: ITT Set
Measure: Median (Full Range); unit: Ratio
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 22 | 20
Ratio | 241 [75 to 528] | 193 [71 to 298]

8. Secondary Outcome: Secondary Efficacy Endpoint -2 : Analysis of Number of Days Without Oxygen Use (Baseline to Day 14)
Description: This secondary efficacy endpoint quantifies the cumulative number of days, from baseline (defined as the start of study intervention or randomization) through Day 14 (inclusive), during which participants did not require supplemental oxygen therapy
Time Frame: Baseline to Day 14
Population: ITT Set
Measure: Median (Full Range); unit: Days
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Days | 0 [0 to 7.2] | 0 [0 to 7.2]

9. Secondary Outcome: Secondary Efficacy Endpoint -3 : Analysis of Number of Days Without Oxygen Use (Baseline to Day 28)
Description: This secondary efficacy endpoint quantifies the cumulative number of days, from baseline (defined as the start of study intervention or randomization) through Day 28 (inclusive), during which participants did not require supplemental oxygen therapy
Time Frame: Baseline to Day 28
Population: ITT Set
Measure: Median (Full Range); unit: Days
Arm/Group | SIR1-365 | Matching placebo
Number analyzed (Participants) | 23 | 19
Days | 1.60 [0 to 27.7] | 3 [0 to 22]

ADVERSE EVENTS:
Time Frame: Baseline to Day 28
Arm/Group | SIR1-365 | Matching placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/23 | 5/19
Other Adverse Events (participants affected / at risk) | 7/23 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIR1-365 (N=23) | Matching placebo (N=19)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Pulmonary embolism
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) — Encephalopathy
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Neck pain
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Respiratory distress
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Acute respiratory failure
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Acute myocardial infarction
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Haemoptysis
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Pneumonia
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Respiratory failure
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIR1-365 (N=23) | Matching placebo (N=19)
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Headache
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) — Burning sensation
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Dizziness
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) — Encephalopathy
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) — Hypoaesthesia
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) — Peripheral sensory neuropathy
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) — Fungal skin infection
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) — Dengue fever
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) — Oral candidiasis
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) — Urinary tract infection
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) — Alanine aminotransferase increased
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) — Aspartate aminotransferase increased
Troponin I increased (Investigations) | 0 (0) | 1 (1) — Troponin I increased
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Hypertension
Hypotension (Vascular disorders) | 1 (1) | 0 (0) — Hypotension
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) — Orthostatic hypotension
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Constipation
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) — Paraesthesia oral
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Hyperkalaemia
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Lactic acidosis
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Acute myocardial infarction
Chest pain (General disorders) | 0 (0) | 1 (1) — Chest pain
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Neck pain
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Pneumonia
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Pulmonary embolism
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Acute respiratory failure
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Haemoptysis
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pulmonary oedema
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Respiratory distress
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Respiratory failure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04622332/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04622332/SAP_001.pdf